CLINICAL TRIAL: NCT02616211
Title: An Integrated Approach to Treating Recurrent Thoracic Carcinomas Resistant to Tyrosine Kinase Inhibitors
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Foundation for Cancer Research (Other)
Responsible Party: Principal Investigator, Jin Jen, M.D., Ph.D., PI, Mayo Clinic
Other Study IDs: 14-002084
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Adenocarcinoma of Lung; Lung Neoplasm; Cancer of Lung; Lung Cancer; Pulmonary Cancer; EGFR Genes; ALK Genes
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the time of recurrence, a minimum of two (2) and a maximum of four (4) tissue cores will be taken through interventional biopsy, ultra sound guided biopsy, surgical resection, or bronchoscopy. Investigators may also collect waste pleural fluid in patients who have a pleurx catheter in place. These biopsies will be collected and individually processed for pathology, gene mutation screening, transcriptome profiling and tumor xenografts.
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients are asked to participate in this study if they have been diagnosed with a thoracic carcinoma which includes lung cancer and have a gene mutation (alteration in the body's genetic instructions) and after undergoing treatment the cancer has come back, progressed, or shown a partial response on standard treatment.

DETAILED DESCRIPTION:
In order to improve the treatment outcome for thoracic carcinomas after they become resistant to targeted therapy, the investigator is using tumor biopsies at the time of recurrence for genomic analysis to identify novel somatic changes in critical genes and gene pathways that can potentially be targeted with therapy. The study team is also creating patient-derived xenografts to test drug efficacy and optimize personalized therapy for each patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Thoracic carcinoma tumors are positive for any targetable genetic alterations
* Have shown partial or no response, progression or recurrence while on or after gene targeted therapy by CT/PET scan
* Tumor is accessible for biopsy or surgery
* Expected life is 6 months or longer.

Exclusion Criteria:

* < 18 years
* Not able to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the Mayo Clinic Rochester
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Identify the number of molecular changes in the recurrent tumor through molecular analysis with gene panels. | 1 Year
  To determine molecular changes in the recurrent tumor, identify the most significant genes and pathways and clinical phenotypes in lung adenocarcinomas resistant to tyrosine kinase inhibitor treatment.
Number of tumorgrafts from biopsies of the recurrent tumor grown and used for drug treatment selection based on genomic signatures. | 1 Year
  Mice will be used to grow tumor xenografts. For subsequent passages, tumors will be implanted through passage mice. The patient-derived xenograft-baring mice will then be used for anti-tumor efficacy studies according to the patient prior therapeutic history and molecular signature of the tumor biopsy.

SECONDARY OUTCOMES:
Recording turn-around-time | 1 year
  Time metrics from biopsy to completion of molecular genetic tests; the time and the success rate of tumorgraft growth in mice as well as the optimal time lapse between initiation treatment to observation of response will be examined. This will aid in the determination of feasibility and opportunities of using patient specific treatment for tumor recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Jen, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials